CLINICAL TRIAL: NCT03234296
Title: Antibiotic Therapy vs. Placebo in the Treatment of Acute Uncomplicated Appendicitis: a Randomized Double-blinded Placebo-controlled Trial - APPAC III Study
Brief Title: Antibiotics vs. Placebo in Acute Uncomplicated Appendicitis
Acronym: APPACIII
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: Tampere University Hospital (Other); Kuopio University Hospital (Other); Oulu University Hospital (Other); Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Paulina Salminen, Primary investigator, Turku University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: APPAC III
Record Dates: First submitted 2017-07-26; First posted 2017-07-31 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Acute Appendicitis
Keywords: uncomplicated acute appendicitis; complicated acute appendicitis; antibiotic therapy; spontaneous resolution
MeSH Terms: conditions — Appendicitis | interventions — Ertapenem; Levofloxacin; Metronidazole

STUDY DESIGN:
Intervention Model Description: Anticipated enrollment delays > three alternate scenarios for sample size calculations, please see prtocol for details.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blinded RCT, no care providers, patients or researchers are aware of the randomised treatment. Separate safety monitoring committee and preplanned interim analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antibiotic treatment (Active Comparator): Ertapenem 1 g x 1 intravenously for 3 days, followed by per oral levofloxacin 500 mg x 1 and metronidazole 500 mg x 3 for 4 days, duration of treatment 7 days.
  Interventions: Drug: Ertapenem
- Placebo (Active Comparator): Intravenous placebo once a day for 3 days, followed by per oral placebo for 4 days with similar p.o. tablets as in the antibiotic group.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ertapenem — Intravenous antibiotic followed by per oral antibiotics
  Other Names: Levofloxacin; Metronidazole
  Arms: Antibiotic treatment
Other: Placebo — Intravenous placebo followed by per oral placebo
  Arms: Placebo

SUMMARY:
Appendicectomy has been the treatment of acute appendicitis for over a hundred years. Appendicectomy, however, includes operative and postoperative risks despite being a "routine" operation. At the same time other similar intra-abdominal infections, such as diverticulitis, are treated with antibiotics. Several studies have proved promising results of the safety and efficiency of antibiotics in the treatment of acute uncomplicated appendicitis. Our previous APPAC study, published in 2015 in the Journal of American Medical Association, also proved promising results with 73% of patients with CT-diagnosed uncomplicated appendicitis treated successfully with antibiotics within one-year follow-up. None of the patients initially treated with antibiotics that later had appendectomy had major complications. The results of the APPAC trial suggest that CT proven uncomplicated acute appendicitis is not a surgical emergency and antibiotic therapy is a safe first-line treatment option. Reducing unnecessary appendectomies has also been shown to lead to significant economic savings.

Already in 1886 Fitz noted that 1/3 of patients in a large series of autopsies from the pre-appendicectomy era had evidence of prior appendices inflammation suggesting spontaneous resolution of acute appendicitis. Acute appendicitis is thought to be similar to acute diverticulitis ("left-sided appendicitis") and this similarity has been shown in epidemiological studies. Recent studies have shown no benefit of antibiotic treatment in the treatment of uncomplicated diverticulitis with outpatient management without antibiotics proving safe and well-functioning.

The aim of this randomised double-blinded study is to compare antibiotic therapy with placebo to evaluate the role of antibiotic therapy in the resolution of CT-diagnosed uncomplicated acute appendicitis.

The hypothesis is that antibiotic therapy is necessary in the treatment of acute uncomplicated appendicitis and that antibiotic therapy is superior to spontaneous resolution (placebo) with the primary endpoint evaluated at ten days after the intervention.

DETAILED DESCRIPTION:
Acute appendicitis is the most common cause of abdominal pain in emergency departments and appendectomy is the most common emergency abdominal surgery. The lifetime risk of acute appendicitis in males is 8.6% and 6.7% in females.In Finland according to Stakes data there were 6 377 appendectomies (3242 in males, 3135 in females, median age 35 years) performed in 2010 with a total number of days in hospital care was 16 111 days and the mean length of hospital stay was three days.

Although acute appendicitis is the most common reason for surgical emergency department visit, its diagnosis still remains challenging. The clinical diagnosis has previously been based on patient history, physical examination and laboratory findings as well as the clinical surgical diagnosis. Several scoring systems have been created to aid in the diagnosis of acute appendicitis18-20, but the accuracy of clinical diagnosis without preoperative imaging is about 76 - 80 % for combined patient groups of males and females.

As acute appendicitis has historically been thought to always progress to perforation requiring emergency appendectomy, high negative appendectomy rates even up to 40 % in some patient populations have been previously accepted as good surgical practice. For the last two decades, the use of dedicated imaging in acute abdomen in general and also in acute appendicitis has led to improved diagnostic accuracy.

Based on large epidemiological studies, it is now known that complicated (perforated) and uncomplicated (non-perforated) appendicitis have followed different epidemiological trends. These unassociated epidemiologic trends suggest different pathophysiology for the two form of appendicitis. The differential diagnosis is essential as patients with an uncomplicated acute appendicitis may not require surgical intervention and might experience even spontaneous resolution without perforation. The majority (approximately 80 %) of acute appendicitis cases are of uncomplicated nature.

Complicated acute appendicitis defined as a finding of a perforation, appendicolith, abscess or a suspicion of a tumor, requires emergency appendectomy with the exception of cases with abscess as they are often managed conservatively.

Appendicolith is a calcified fecal concretion in the appendix resulting in internal luminal obstruction and it is the most common form of complicated acute appendicitis. In the first randomized study by Vons et al. comparing operative treatment and antibiotic therapy using CT as a diagnostic inclusion criterion, the presence of an appendicolith in preoperative CT scan was the only factor that significantly increased the risk of complicated appendicitis and it was also the only factor associated with the failure of antibiotic therapy for acute appendicitis. Indeed, if Vons et al had excluded the patients with an appendicolith from their analysis, no significant difference in the incidence of post-intervention peritonitis between the treatment groups would have been noticed in their study.

CT imaging is the primary imaging modality and the golden standard in the diagnosis of acute appendicitis as it establishes the diagnosis with almost perfect diagnostic accuracy. The advantages of CT imaging are high accuracy, availability, ease of performance and interpretation, and that it is rarely affected by bowel gas, severe abdominal pain or extreme body habitus. The main disadvantage of CT is exposure to radiation.

The increased use of preoperative CT imaging has been evaluated thoroughly by evaluating its impact on the negative appendectomy rate reducing the number of unnecessary appendectomies. In 2010, a mandatory imaging guideline for suspected acute appendicitis was implemented in the Netherlands. After implementation the negative appendectomy rate dropped significantly from 23 % to 6 % (p<0.001) reducing the surgical complication rate from 20% to 14 % and resulting in average cost-per-patient decrease by 594€.

The favorable diagnostic performance of CT imaging has encouraged optimization of the protocol to minimize exposure to radiation through the development of low-dose CT protocols. Low-dose protocols balance with as low as reasonably achievable-principle while maintaining diagnostic accuracy. However, low-dose protocols with intravenous contrast are still not implemented in routine clinical practice. These protocols require more advanced optimization and validation because of the wider need for contrast enhanced assessment. Kim et al showed that contrast enhanced low-dose CT (median radiation dose 116 mmGy in dose-length product) was not inferior to standard-dose contrast enhanced CT (median radiation dose 521 mmGy), with negative appendectomy rates of 3.5% and 3.2% respectively and no statistical significance in appendiceal perforation rates or patients requiring additional imaging.

The investigators have performed a prospective observational study (OPTICAP trial, NCT02533869, Ethical committee of Turku University Hospital approval) in order to optimize a low-dose CT scan for both diagnosing acute appendicitis and to differentiate uncomplicated acute appendicitis from a complicated acute appendicitis. In this study, phantom imaging with 15 different imaging protocols were performed aiming to minimize radiation with optimal diagnostic accuracy. The phantom protocols were assessed by blinded evaluation of two gastrointestinal radiologists and the two best performing protocols were chosen for the clinical phase. The clinical evaluation included performing both of these imaging protocols for patients with suspected uncomplicated acute appendicitis evaluated by a senior digestive surgeon. All of the enrolled patients underwent laparoscopic appendectomy to evaluate the sensitivity and specificity of the imaging protocols. The two most optimal imaging protocol were selected for use in the APPAC III trial; one low-dose CT protocol for patients with BMI> 30 and one optimised standard CT for patients with BMI exceeding 30.

For over a century appendectomy has been the standard treatment for all patients with acute appendicitis. However, the results of our APPAC trial have now shown that the majority (73%) of patients with uncomplicated acute appendicitis were successfully treated with antibiotics alone. We also showed that none of the patients treated initially with antibiotics and later undergoing appendectomy had major complications or increased morbidity defining antibiotic therapy as a safe first-line treatment. Patients with a complicated acute appendicitis require emergency appendectomy and early identification of these patients is of vital importance. Laparoscopic appendectomy has become the golden standard for appendectomy providing lower morbidity and faster recovery compared with open appendectomy. For patients with uncomplicated acute appendicitis, the time has come to evaluate abandoning routine appendectomy and evaluating the optimal use of antibiotic therapy.

Emergency appendectomy was first advocated because of the very high mortality of perforated appendicitis combined with the assumption of the natural course of acute appendicitis evolving always to perforated disease. This was first reported in 1886 by Reginald Fitz, who initially originated the term appendicitis and identified appendix as a cause for right lower quadrant infections. Fitz also noted that one-third of patients in a large autopsy series from the pre-appendectomy era had evidence of prior appendiceal inflammation suggesting spontaneous resolution of acute appendicitis.

Acute appendicitis is similar to acute diverticulitis ("left-sided appendicitis") and this similarity has been shown in epidemiological studies suggesting a common underlying pathogenesis. There is one multicenter randomized trial, one population-based study, one case-control study and one prospective observational study that have shown no benefit of antibiotic therapy in uncomplicated acute diverticulitis. The reported complication rates in these studies is low (approximately 2 %) and even outpatient management without antibiotics in acute uncomplicated diverticulitis has been shown to be feasible, well-functioning and safe. The APPAC III trial will first recruit 3-5 pilot patients in order to finalise the hospital pharmacy procedures in practice.

The aim of the APPAC III study is to compare antibiotic therapy with placebo in the treatment of uncomplicated acute appendicitis to evaluate the role of antibiotic therapy in the resolution of acute uncomplicated appendicitis. The study hypothesis is that antibiotic therapy is necessary in the treatment of acute uncomplicated and that antibiotic therapy is superior to spontaneous resolution (placebo) with the primary endpoint evaluated at ten days after the intervention.

Sample size calculations were based on one-sided Pearson's χ2 -test for two proportions. Sample size was calculated from an estimated success rate of 94% during the hospitalization in antibiotic group 7. A decrease of 15 percentage points in success rate is considered clinically important difference leading to estimated 79% success rate in placebo group. We estimated that to detect a 15 percentage points difference (antibiotics - placebo) between groups with a power of 0.8 (1-β) and one-sided significance level (α) of 0.05 64 patients per group is needed. Before the trial initiation, 3-5 pilot patients will be recruited in order to finalize the hospital pharmacy procedures and drug delivery in clinical practice. Based on the pilot study enrollment speed and the recognized challenges in conducting trial, in real-life emergency setting we need to take into account the anticipated enrolment delays to assure the completion of this trial within reasonable time. These challenges consisting of emergency surgery patient enrolment dependent on hospital pharmacy services available only during standard working hours, the requirement for senior surgeon enrolment and the discrepancy between the admission hours of appendicitis patients and hospital pharmacy working hours mandated us to create three scenarios for study power analysis and the number of patients to be enrolled.

In scenario A, a decrease of 15 percentage points in success rate is considered clinically important difference leading to estimated 79% success rate in placebo group. We estimated that to detect a 15-percentage points difference (antibiotics - placebo) between groups 64 patients per group is needed. With an estimated dropout rate of 10% total of 142 patients, 71 patients per group will be enrolled in the study. In scenario B, clinically important difference is 20 percentage points, estimated success rate in placebo group is 74% and to detect this difference 41 patients per group is needed. With an estimated dropout rate of 10% total of 92 patients, 46 patients per group will be enrolled in the study. In scenario C, clinically important difference is 25 percentage points, estimated success rate in placebo group is 69% and to detect this difference 29 patients per group is needed. With an estimated dropout rate of 10% total of 64 patients, 32 patients per group will be enrolled in the study. Targeted minimum sample size per study hospital will be 10 patients. One-sided test will be used as our hypothesis is that antibiotic treatment is more effective treatment than placebo. Sample size calculations were performed using Power procedure in SAS System for Windows, Version 9.4 (SAS Institute Inc., Cary, NC).

On April 1st, 2019, a study committee consisting of the outside safety monitoring committee and the core research group will assess which one of these scenarios is most feasible based on patient enrolment with plan A being the target scenario. Active recruitment at this point will be continued until a decision is made on the clinically realistic enrolment scenario. The date of evaluation is set exactly one year after the last study hospital has initiated enrolment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-60 years
* CT confirmed uncomplicated acute appendicitis
* Ability to give informed consent

Exclusion Criteria:

* Age under 18 or over 60 years
* Pregnancy or lactation
* Allergy to contrast media or iodine
* Allergy or contraindication to antibiotic therapy
* Metformin medication
* Renal insufficiency
* Severe systemic illness (for example malignancy, medical condition requiring immunosuppressant medication)
* Complicated acute appendicitis confirmed by CT scan
* Inability to cooperate or give informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 147 (Estimated)
Dates: Start 2017-08-09 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2029-08-30 (Estimated)

PRIMARY OUTCOMES:
Success of the randomized treatment | 10 days after treatment initiation
  Resolution of acute appendicitis with study group treatment resulting in discharge from the hospital without the need for surgical intervention and treatment efficacy evaluated at ten days after initiation of the randomized treatment.

SECONDARY OUTCOMES:
Late recurrence of appendicitis | 10 years
  Late recurrence of acute appendicitis after study treatment defined as clear clinical suspicion of acute appendicitis evaluated at follow-up of one, three, five and ten years
Post-intervention complications | 10 years
  Complications according to the Clavien-Dindo classification
Hospital stay | 1 month
  Duration of hospital stay in days
VAS score (visual analogue score) | 10 years
  Pain as defied by the VAS pain score
Sick leave | 1 month
  Duration of sick leave
Treatment costs | 10 years
  Costs resulting from laboratory costs, imaging costs, treatments costs, hospital stay, and treatment of complications and possible operative treatment

CONTACTS AND LOCATIONS:
Overall Officials: Paulina Salminen, MD,PhD, Principal Investigator — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Salminen P, Sippola S, Haijanen J, Nordstrom P, Rantanen T, Rautio T, Sallinen V, Loyttyniemi E, Hurme S, Tammilehto V, Laukkarinen J, Savolainen H, Merilainen S, Leppaniemi A, Gronroos J. Antibiotics versus placebo in adults with CT-confirmed uncomplicated acute appendicitis (APPAC III): randomized double-blind superiority trial. Br J Surg. 2022 May 16;109(6):503-509. doi: 10.1093/bjs/znac086. PMID 35576384
- [Derived] Sippola S, Gronroos J, Sallinen V, Rautio T, Nordstrom P, Rantanen T, Hurme S, Leppaniemi A, Merilainen S, Laukkarinen J, Savolainen H, Virtanen J, Salminen P. A randomised placebo-controlled double-blind multicentre trial comparing antibiotic therapy with placebo in the treatment of uncomplicated acute appendicitis: APPAC III trial study protocol. BMJ Open. 2018 Nov 3;8(11):e023623. doi: 10.1136/bmjopen-2018-023623. PMID 30391919